CLINICAL TRIAL: NCT06518967
Title: Analytical Performance Study of the Handheld Device Single-Molecule with a Large Transistor (SiMoT) for the Near-patient Testing of Biological Samples
Brief Title: Performance Study with the SiMoT System for in Vitro Diagnostic Tests
Status: Active, not recruiting | Type: Observational
Sponsor: Centro di Innovazione Regionale in Single Molecule Digital Assay (Other)
Responsible Party: Sponsor
Other Study IDs: SiMoT-01
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Non-interventional Analytical Performance Study on Left-over Samples

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open: Test analysis perfomed in open to train the artificial intelligence algorithm.
  Interventions: Diagnostic Test: analytical performance study
- Blind: Test analysis performed in blind to minimize biases when evaluating the predictive performance of the IVD under investigation.
  Interventions: Diagnostic Test: analytical performance study

INTERVENTIONS:
Diagnostic Test: analytical performance study — analytical performance study on left-over samples with the SiMoT IVD system for in vitro diagnostic tests

SUMMARY:
Advanced and performing technologies able to analyze specific biomarkers for the diagnosis, prognosis and prediction as well as for the monitoring, the personalized care and the evaluation of the therapeutic response to pathologies, is currently considered extremely relevant. Such technologies work only if molecular markers specific for a given pathology have been already validated. This approach is considered of strategic importance for the health and well-being of citizens as well as for the sustainability of public spending. Often, however, the analysis of the markers is carried out on tissues or fluids of the organs involved, being hence quite invasive procedures. In this scenario, it is strategic to develop devices and platforms that allow the analysis of markers in a minimally invasive or non-invasive way, through the analysis of peripheral biological fluids, such as blood or urine. The goal is to provide clinicians with the attacker's advantage against a plethora of progressive diseases by mass-screening individuals who are affected by a disease long before symptoms appear or to allow the identification of those patients who have a high probability of recurring or responding to target-oriented pharmacological approaches. This study pertains to the definition of the analytical performance of the Single-Sensor Single-Molecule with a large Transistor (SiMoT) device. In the context of the present performance study, the IVD SiMoT system will be equipped with an accessory-cartridge developed and produced without any diagnostic purpose but only to verify the analytical performance of the SiMoT system, in the detection of exogenous biochemical molecules suitably selected to act as markers of interest.

DETAILED DESCRIPTION:
Advanced and performing technologies able to analyze specific biomarkers for the diagnosis, prognosis and prediction as well as for the monitoring, the personalized care and the evaluation of the therapeutic response to pathologies, is currently considered extremely relevant. Such technologies work only if molecular markers specific for a given pathology have been already validated. This approach is considered of strategic importance for the health and well-being of citizens as well as for the sustainability of public spending. Among the pathologies that will increasingly be monitored and treated thanks to enabling technologies for precision medicine, tumors are certainly of particular importance. Often, however, the analysis of the markers is carried out on tissues or fluids of the organs involved, being hence quite invasive procedures. In this scenario, it is strategic to develop devices and platforms that allow the analysis of markers in a minimally invasive or non-invasive way, through the analysis of peripheral biological fluids, such as blood or urine. The goal is to provide clinicians with the attacker's advantage against a plethora of progressive diseases by mass-screening individuals who are affected by a disease long before symptoms appear or to allow the identification of those patients who have a high probability of recurring or responding to target-oriented pharmacological approaches.

This study pertains to the definition of the analytical performance of the Single-Sensor Single-Molecule with a large Transistor (SiMoT) device. The SiMoT device is an in vitro diagnostic - IVD system (REGULATION (EU) 2017/746, IVDR Art. 2, point 2) that performs decentralized analyses (near-patient testing, such as, for example, patient's home, emergency unit, ambulance) composed of a palm reader completed by machine-learning / artificial-intelligence software. The system works through an accessory (IVDR Art. 2, point 4) represented by a disposable cartridge, which determines the specific diagnostic application based on the molecular markers detected by the accessory. In the context of the present performance study, the IVD SiMoT system will be equipped with an accessory-cartridge developed and produced without any diagnostic purpose but only to verify the analytical performance of the SiMoT system, in the detection of exogenous biochemical molecules suitably selected to act as markers of interest.

The present performance study aims to verify the qualitative detection (on/off) of target molecules (both proteins and nucleic acids) with a single molecule threshold in 0.1 mL (10^-20 M). The threshold is established by the limit of identification (LOI).

Analytical performance will be evaluated according to standard statistical approaches such as: analytical sensitivity, analytical specificity, trueness (bias), precision (repeatability and reproducibility), accuracy (resulting from trueness and precision), limits of detection and identification, measurement range, possible linearity, threshold values, including the determination of appropriate criteria for the collection and handling of samples and the control of known endogenous and exogenous interferences, cross reactions.

Risk evaluation (Risk-to-Benefits rationale) There are no identifiable physical, psychic and/or social risks for the patients enrolled in the study directly deriving from the procedures that will be followed for the enrollment and collection of the related data.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent and personal data handling consent signed by the subject;
* > 18 years of age
* presence of neoplastic or suspected neoplastic pathology at the time of sample collection

Exclusion Criteria:

* < 18 years of age
* Participation in a clinical trial with an investigational drug or a medical device within the 30 days preceding and during the present investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves around 50 patients with solid tumors who will come to the Gynecological Oncologic Clinic at IRCCS Giovanni Paolo II Cancer Institute and who are prescribed for pre-hospitalization procedures as per standard clinical practice at the investigational site.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the analytical performance in plasma, serum, and urine samples supplemented with non-endogenous molecules (three proteins and two nucleotide sequences) of the SiMoT handheld device | December 2024
  Qualitative detection of specific marker at single molecule level

SECONDARY OUTCOMES:
Duration of analytical analysis performance | December 2024
  To define the time to obtain the test result (time-to-result) for a complete analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Tumori Giovanni Paolo II, Gynecological Oncologic Clinic, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No